CLINICAL TRIAL: NCT06342986
Title: Intraperitoneal FT536 in Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023LS185; P01CA111412 (NIH)
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Gynecologic Cancer; Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — fludarabine

STUDY DESIGN:
Intervention Model Description: A minimum of 28 days must separate each Dose Cohort. A minimum of 30 days must separate the 1st and 2nd patient. All patients are assessed for Dose Limiting Toxicity (DLT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Cohort -1: IP FT536 monotherapy 3 x 10^6 cells/dose (Experimental): FT536 is an allogeneic natural killer (NK)-cell immunotherapy produced from a clonal master human induced pluripotent stem cell (iPSC) line with the following engineered elements: a) deletion of the gene encoding CD38 (i.e., CD38 knockout) and expression of the MICA and MICB (MICA/B) chimeric antigen receptor (CAR); b) high-affinity, non-cleavable CD16 receptor; and c) interleukin (IL)-15/IL-15 receptor alpha fusion protein. Participants will receive doses on Day 1, Day 4 and day 8.
  Interventions: Drug: FT536; Drug: Fludarabine; Drug: CY
- Dose Cohort 1: IP FT536 monotherapy 1 x 10^8 cells/dose (Experimental): FT536 is an allogeneic natural killer (NK)-cell immunotherapy produced from a clonal master human induced pluripotent stem cell (iPSC) line with the following engineered elements: a) deletion of the gene encoding CD38 (i.e., CD38 knockout) and expression of the MICA and MICB (MICA/B) chimeric antigen receptor (CAR); b) high-affinity, non-cleavable CD16 receptor; and c) interleukin (IL)-15/IL-15 receptor alpha fusion protein. Participants will receive doses on Day 1, Day 4 and day 8.
  Interventions: Drug: FT536; Drug: Fludarabine; Drug: CY
- Dose Cohort 2: IP FT536 monotherapy 3 x 10^8 cells/dose (Experimental): FT536 is an allogeneic natural killer (NK)-cell immunotherapy produced from a clonal master human induced pluripotent stem cell (iPSC) line with the following engineered elements: a) deletion of the gene encoding CD38 (i.e., CD38 knockout) and expression of the MICA and MICB (MICA/B) chimeric antigen receptor (CAR); b) high-affinity, non-cleavable CD16 receptor; and c) interleukin (IL)-15/IL-15 receptor alpha fusion protein. Participants will receive doses on Day 1, Day 4 and day 8.
  Interventions: Drug: FT536; Drug: Fludarabine; Drug: CY
- Dose Cohort 3: IP FT536 monotherapy 1 x 10^9 cells/dose (Experimental): FT536 is an allogeneic natural killer (NK)-cell immunotherapy produced from a clonal master human induced pluripotent stem cell (iPSC) line with the following engineered elements: a) deletion of the gene encoding CD38 (i.e., CD38 knockout) and expression of the MICA and MICB (MICA/B) chimeric antigen receptor (CAR); b) high-affinity, non-cleavable CD16 receptor; and c) interleukin (IL)-15/IL-15 receptor alpha fusion protein. Participants will receive doses on Day 1, Day 4 and day 8.
  Interventions: Drug: FT536; Drug: Fludarabine; Drug: CY

INTERVENTIONS:
Drug: FT536 — FT536 is an allogeneic natural killer (NK)-cell immunotherapy produced from a clonal master humaninduced pluripotent stem cell (iPSC) line.
Drug: Fludarabine — Fludarabine 25 mg/m2 IV given on day -5. Given consecutively with CY.
Drug: CY — CY 300 mg/m2 IV given on day -4. Given consecutively with Fludarabine.

SUMMARY:
This is a single center Phase I clinical trial of FT536 administered intraperitoneally (IP) 3 times a week for one week for the treatment of recurrent gynecologic cancers. A short course of outpatient lymphodepleting chemotherapy is given prior to the first dose of FT536 to promote adoptive transfer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian cancer, fallopian tube, or primary peritoneal cancer meeting one of the following minimal prior treatment requirements (no limit to the maximum number of prior treatments).
* Must have received prior bevacizumab.
* In the presence of a BRCA mutation, must have received a prior PARP inhibitor.
* Adequate organ function within 14 days (28 days for pulmonary and cardiac) of study treatment (CY/Flu) start
* Agrees to the placement of an intraperitoneal catheter before the 1st dose of study directed drug (chemotherapy) and remains in place through Day 36 or longer if retreatment is planned. Refer to Section 6.4 if catheter cannot be successfully placed.
* Agrees to undergo a tumor biopsy if feasible at the time the catheter is placed and removed - Accessible tumor for biopsy is not required for eligibility
* Must agree to and sign the consent for the companion Long-Term Follow-Up study (CPRC# 2021LS077) to fulfill the FDA recommended 15 years of followup for a genetically modified cell product.

Exclusion Criteria:

* Pregnant or breastfeeding or planning on becoming pregnant in the next 6 months. If of childbearing potential (have a uterus and ovaries) and engaged in heterosexual intercourse, must have a negative pregnancy test (serum or urine) within 14 days before the 1st CY/Flu. Patient must agree to use highly effective method of birth control from the screening visit until at least 12 months after the final dose of CY, or at least 4 months after the final dose of FT536, whichever is longer.
* Currently receiving or likely to require systemic immunosuppressive therapy (e.g., prednisone >5 mg daily) for any reason from Day -5 to 14 days after the last FT536 infusion) with the exception of corticosteroids as a pre-medication per institutional standard of care - topical and inhaled steroids are permitted.
* Active autoimmune disease requiring systemic immunosuppressive therapy.
* History of severe asthma and currently on chronic systemic medications.
* Uncontrolled bacterial, fungal or viral infections with progression of clinical symptoms despite therapy.
* Receipt of any biological therapy, chemotherapy, or radiation therapy (except palliative RT), within 2 weeks prior to the first dose of FT536 or five half-lives, whichever is shorter; or any investigational agent within 28 days prior to the first dose of FT536.
* Live vaccine within 6 weeks prior to start of lympho-conditioning.
* Known allergy to the following FT536 components: albumin (human) or dimethyl sulfoxide (DMSO).
* Prior enoblituzumab.
* Non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions in the 2-year period leading up to study enrollment. (Refer to Section 5.1.8 regarding history of brain metastases.)
* Known history of HIV positivity or active hepatitis C or B - chronic asymptomatic viral hepatitis is allowed.
* Presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to patient.
* Any medical condition or clinical laboratory abnormality that, per investigator judgement, precludes safe participation in and completion of the study or that could affect compliance with protocol conduct or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 1 year

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 months
Overall survival (OS) | 6 months
Overall survival (OS) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No